CLINICAL TRIAL: NCT07401069
Title: The Effect of Homemade Herbal Mouthwash Versus Chlorhexidine on Plaque Accumulation in Gingivitis. A Randomized Clinical Trial.
Brief Title: Homemade Herbal Mouthwash in Gingivitis. A Randomized Clinical Trial.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayat Gamal-AbdelNaser, PI, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACU-Per3
Record Dates: First submitted 2026-02-01; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine mouthwash (Active Comparator)
  Interventions: Drug: Chlorhexidine 0,12%
- Herbal Homemade Mouthwash (Experimental)
  Interventions: Drug: herbal Mouthwash

INTERVENTIONS:
Drug: Chlorhexidine 0,12% — chlorhexidine 0.12% mouthwash twice daily for 7 days
  Arms: Chlorhexidine mouthwash
Drug: herbal Mouthwash — Mouthwash made at home by boiling herbs in water and then saving the solution in a tightly closed container for daily use for 7 days
  Arms: Herbal Homemade Mouthwash

SUMMARY:
Gingivitis is a very common oral disease that may progress to the more destructive periodontitis if not treated. As oral plaque is a key player in gingivitis, plaque control by professional scaling and oral hygiene measures represents the main line of treatment.

Among the oral hygiene measures, using chlorhexidine mouthwash is considered the gold standard in mouthwashes. However, due to its side effects, a safer and more acceptable mouthwash is needed. Therefore, this study proposes mouthwashes made of infusion of natural herbs as an alternative.

ELIGIBILITY:
Inclusion Criteria:

* Plaque-induced gingivitis.

Exclusion Criteria:

* Medically compromised.
* History of medications.
* Pregnant females.
* Periapical involvement in teeth.
* History of periodontal surgery.
* If gingivitis was due to local factor.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
plaque index (O'Leary et al., 1972) | 7 days
  Plaque accumulation is tested on teeth with a probe. Number of sites having plaque accumulation will be divided by the total number of dental sites to get percentage of plaque accumulation.

SECONDARY OUTCOMES:
Bleeding on probing | 7 days
  Bleeding on probing is tested on teeth with a periodontal probe. Number of sites showing bleeding will be divided by the total number of dental sites to get percentage of bleeding on probing.
Changes in clinical signs of inflammation (Armitage, 2004) | 7 days
  Results will be in the form of (Yes/No); indicating if the gingival clinical condition (color and contour) was improved or not
Bleeding on brushing | 7 days
  Evaluation of extent of daily bleeding on brushing using VAS.
Patient's acceptance of the mouthwash | 7 days
  questionnaire